CLINICAL TRIAL: NCT01840449
Title: Non-interventional, Observational Study to Evaluate Common Therapeutic Algorithms and Possible Predictive Parameters for Somatuline Autogel® (ATG) Treatment in Subjects With Either Acromegaly or Neuroendocrine Tumours (NET)
Brief Title: Somatuline Predictive Factors in Acromegaly and NET
Acronym: SOPRANo
Status: Completed | Type: Observational
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: A-94-52030-240
Record Dates: First submitted 2013-04-23; First posted 2013-04-25 (Estimated); Last update posted 2019-01-14 (Actual); Status verified 2019-01

CONDITIONS: Acromegaly; Neuroendocrine Tumours
MeSH Terms: conditions — Acromegaly; Neuroendocrine Tumors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Neuroendocrine Tumours: The subject will receive treatment as prescribed by the investigator and in accordance with the current recommendations, routine practice and local regulations.
  Interventions: Drug: Somatuline Autogel® 60, 90 or 120 mg
- Acromegaly: The subject will receive treatment as prescribed by the investigator and in accordance with the current recommendations, routine practice and local regulations.
  Interventions: Drug: Somatuline Autogel® 60, 90 or 120 mg

INTERVENTIONS:
Drug: Somatuline Autogel® 60, 90 or 120 mg

SUMMARY:
The aim of the study is to identify predictive factors for the response to Lanreotide treatment in Acromegaly as well as in Neuroendocrine Tumours.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent (also mandatory in case of retrospective documentation of subject data)
* Diagnosis of acromegaly or NET with the intention to be treated with ATG or already on treatment with ATG

Exclusion Criteria:

* The subject has already been included in this study
* Participation in an interventional trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Clinics and private practitioners who treat acromegaly and/or NET subjects with Somatuline Autogel® 60, 90 or 120 mg.
Sampling Method: Non-Probability Sample
Enrollment: 156 (Actual)
Dates: Start 2012-06; Primary Completion 2016-07 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Change in biochemical markers (Growth Hormone [GH] & Insulin-like Growth Factor 1 [IGF-1] in acromegaly subjects and Chromogranin A [CgA] in NET subjects) | Baseline and 1 year

SECONDARY OUTCOMES:
Change in biochemical markers (Growth Hormone [GH] & Insulin-like Growth Factor 1 [IGF-1] in acromegaly subjects and Chromogranin A [CgA] in NET subjects) | Baseline and 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (3):
- University Hospital of Vienna, Vienna, Austria
- ENDOC, Hamburg, Germany
- University Hospital Basel, Basel, Switzerland

REFERENCES:
- [Derived] Rinke A, Maintz C, Muller L, Weber MM, Lahner H, Pavel M, Saeger W, Houchard A, Ungewiss H, Petersenn S. Multicenter, Observational Study of Lanreotide Autogel for the Treatment of Patients with Neuroendocrine Tumors in Routine Clinical Practice in Germany and Austria. Exp Clin Endocrinol Diabetes. 2021 Jul;129(7):500-509. doi: 10.1055/a-1342-2755. Epub 2021 Jul 22. PMID 34293802